CLINICAL TRIAL: NCT01024608
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Phase 3 Study to Assess the Efficacy and Safety of Beclomethasone Dipropionate Hydrofluoroalkane (BDP HFA) Nasal Aerosol in Subjects 12 Years of Age and Older With SAR
Brief Title: Study in Adult and Adolescent Subjects With Seasonal Allergic Rhinitis (SAR)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BDP-AR-301
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Results first posted 2012-05-23 (Estimated); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Seasonal Allergic Rhinitis; Hay Fever
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Beclomethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BDP HFA 320 µg/day (Experimental): During the 2-week double-blind Treatment Period participants self-administered 4 actuations (two per nostril) of 80 µg BDP HFA once daily each morning.
  Interventions: Drug: Beclomethasone dipropionate
- Placebo (Placebo Comparator): During the 2-week double-blind Treatment Period participants self-administered four actuations (two per nostril) of placebo HFA once daily each morning.
  Interventions: Drug: Placebo Nasal Aerosol

INTERVENTIONS:
Drug: Beclomethasone dipropionate — Total daily dose of 320 micrograms per day of beclomethasone dipropionate (BDP) hydrofluoroalkane (HFA) applied as a nasal aerosol each morning for two weeks.
  Other Names: QNASL(TM)
  Arms: BDP HFA 320 µg/day
Drug: Placebo Nasal Aerosol — Placebo nasal aerosol administered each morning for two weeks.
  Arms: Placebo

SUMMARY:
The purpose of the study is to assess the efficacy and safety of an investigational nasal aerosol compared with placebo nasal aerosol in the treatment of seasonal allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* Male or female subjects 12 years of age or older
* Documented history of season allergic rhinitis to mountain cedar pollen
* General good health
* Other criteria apply

Exclusion Criteria:

* History of physical findings of nasal pathology (within 60 days prior to screening visit)
* Participation in any investigational drug study 30 days preceding screening visit
* History of respiratory infection/disorder with 14 days preceding screening visit
* Use of any prohibited concomitant medications
* Other criteria apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2009-12-31 (Actual); Primary Completion 2010-02-28 (Actual); Study Completion 2010-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sudeesh Tantry, Ph.D., Study Director — Teva Branded
Locations (4):
- United States (4):
  - Teva Clinical Trial Site, Austin, Texas
  - Teva Clinical Trial Site, New Braunfels, Texas
  - Teva Clinical Trial Site, San Antonio, Texas
  - Teva Clinical Trial Site, Waco, Texas

REFERENCES:
- [Result] Van Bavel J, Ratner PH, Amar NJ, Hampel FC, Melchior A, Dunbar SA, Tantry SK and Dorinsky PM (2011). BDP HFA Nasal Aerosol 320 μg Once Daily Effectively Improves Ocular Symptoms Associated With Seasonal Allergic Rhinitis. Ann Allergy Asthma Immunol. 107(11):A118.
- [Result] Van Bavel J, Dorinsky PM, Melchior A, Dunbar SA, and Tantry SK (2011). Nasal Symptom Relief and Improvement in Health-Related Quality of Life Following Treatment with BDP HFA Nasal Aerosol (320 mcg Once Daily) in Subjects with Seasonal Allergic Rhinitis. Allergy Asthma Proc. 32(4):330.
- [Result] Van Bavel J, Hampel, FC, Ratner PH, Melchior A, Dunbar SA, Tantry SK and Dorinsky PM (2011). BDP HFA Nasal Aerosol Effectively Improves Nasal Symptom Relief and Health-Related Quality of Life (QOL) in Subjects with Seasonal Allergic Rhinitis (SAR). J Allergy Clin Immunol. 127(2):201.
- [Result] Van Bavel J, Amar NJ, Melchior A, Dunbar SA, Tantry SK and Dorinsky PM (2010).BDP HFA Nasal Aerosol, 320 mcg Once Daily, is Safe and Effective in the Treatment of Nasal Symptoms Associated with Seasonal Allergic Rhinitis (SAR). Ann Allergy Asthma Immunol. 105(5):121.
- [Derived] van Bavel JH, Ratner PH, Amar NJ, Hampel FC Jr, Melchior A, Dunbar SA, Dorinsky PM, Tantry SK. Efficacy and safety of once-daily treatment with beclomethasone dipropionate nasal aerosol in subjects with seasonal allergic rhinitis. Allergy Asthma Proc. 2012 Sep-Oct;33(5):386-96. doi: 10.2500/aap.2012.33.3593. PMID 23026180

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 484 patients were screened and 463 patients were enrolled in the study and participated in the Run-in Period. Of the 463 enrolled patients, 340 were randomized to study treatment.
Pre-assignment Details: During the 7 to 10 day Run-in Period, participants self-administered a single-blind placebo nasal aerosol once daily in the morning and assessed and recorded their seasonal rhinitis symptoms twice daily to determine eligibility for randomization.
Groups:
- BDP HFA 320 µg/Day: During the 2-week double-blind Treatment Period participants self-administered 4 actuations (two per nostril) of 80 µg beclomethasone dipropionate (BDP) hydrofluoroalkane (HFA) once daily each morning.
Period: Overall Study
Arm/Group | BDP HFA 320 µg/Day | Placebo
Started | 169 | 171
Intent to Treat Population | 167 (Participants who received at least 1 dose of study drug and had at least 1 post-baseline assessment) | 171 (Participants who received at least 1 dose of study drug and had at least 1 post-baseline assessment)
Safety Population | 167 (Participants who received at least 1 dose of study drug) | 171 (Participants who received at least 1 dose of study drug)
Completed | 165 | 167
Not Completed | 4 | 4
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 0 | 3
Not completed — Never received study treatment | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BDP HFA 320 µg/Day | Placebo | Total
Number analyzed (Participants) | 167 | 171 | 338
Age, Continuous [Mean (Standard Deviation); unit: years] — Demographic data are provided for the Intent to Treat population.
  years | 39.3 (13.4) | 38.0 (13.3) | 38.6 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 97 | 210
  Male | 54 | 74 | 128
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 52 | 49 | 101
  Not Hispanic or Latino | 115 | 122 | 237
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants] — A participant may select more than one race type.
  participants
    American Indian or Alaska Native | 1 | 1 | 2
    Asian | 3 | 3 | 6
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Black or African American | 23 | 26 | 49
    White | 142 | 142 | 284

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Subject-Reported AM and PM Reflective Total Nasal Symptom Score (rTNSS) Over the Two-week Treatment Period
Description: Participants recorded the severity of their nasal symptoms (sneezing, runny nose, nasal itching and nasal congestion) over the past 12 hours (prior to the assessment) twice daily (AM and PM) using the following scale:
  0=absent (no sign/symptom present); 1=mild (sign/symptom present, easily tolerated); 2=moderate (definite awareness of sign/symptom, bothersome but tolerable); 3=severe (hard to tolerate, interfere with daily activities and/or sleeping).
  The rTNSS (sum of 4 symptom scores) ranges from 0 to 12 (worst symptoms). A negative change from baseline score indicates symptom improvement.
Time Frame: Baseline (Days -3 to 0), and Days 1-15
Population: Intent to treat population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BDP HFA 320 µg/Day | Placebo
Number analyzed (Participants) | 167 | 171
units on a scale | -2.0 (0.16) | -1.0 (0.15)
Statistical Analysis 1: Comparison: BDP HFA 320 µg/Day vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — A priori threshold for statistical significance is p<0.05; Repeated measures ANCOVA included covariate adjustment for baseline, day, treatment, and the treatment by day interaction; LS mean treatment diff from placebo = -0.91, 95% CI 2-sided [-1.3 to -0.5]

2. Secondary Outcome: Change From Baseline in Average Subject-Reported AM and PM Instantaneous Total Nasal Symptom Score (iTNSS) Over the Two-week Treatment Period
Description: Participants recorded the severity of their nasal symptoms (sneezing, runny nose, nasal itching and nasal congestion) over the past 10 minutes (prior to the assessment) twice daily (AM and PM) using the following scale:
  0=absent (no sign/symptom present); 1=mild (sign/symptom present, easily tolerated); 2=moderate (definite awareness of sign/symptom, bothersome but tolerable); 3=severe (hard to tolerate, interfere with daily activities).
  The iTNSS (sum of the 4 symptom scores) ranges from 0 to 12 (worst symptoms). A negative change from baseline score indicates symptom improvement.
Time Frame: Baseline (Days -3 to 0), and Days 1-15
Population: Intent to treat population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BDP HFA 320 µg/Day | Placebo
Number analyzed (Participants) | 167 | 171
units on a scale | -1.7 (0.15) | -0.8 (0.15)
Statistical Analysis 1: Comparison: BDP HFA 320 µg/Day vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — A priori threshold for statistical significance is p<0.05; The repeated measures ANCOVA included covariate adjustment for baseline, day, treatment, and the treatment by day interaction; LS mean treatment diff from placebo = -0.92, 95% CI 2-sided [-1.3 to -0.5]

3. Secondary Outcome: Change From Baseline at Week 2 in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) in Participants With Impaired Quality of Life at Baseline
Description: The adult RQLQ has 28 questions in 7 domains. Participants were asked to recall their experiences during the previous week and to give their responses on a 7-point scale (0 = Not Troubled to 6 = Extremely Troubled) for the domains of activities, sleep, non-nose/eye symptoms, practical problems, nasal symptoms, and eye symptoms. The domain of 'emotional' utilized a separate scale (0 = None of the time to 6 = All of the time). The overall RQLQ score is the mean of all 28 responses. Week 2 scores were compared to baseline scores. A negative change from baseline score indicates improvement.
Time Frame: Day 0 (Baseline), Day 15
Population: The RQLQ population, subset of ITT population, included only those participants over the age of 18 years (fluent in English) with an impaired quality of life at Baseline as defined by a RQLQ score at Day 0 of 3.0 or greater.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BDP HFA 320 µg/Day | Placebo
Number analyzed (Participants) | 129 | 121
units on a scale | -1.2 (0.12) | -0.8 (0.12)
Statistical Analysis 1: Comparison: BDP HFA 320 µg/Day vs Placebo; Test type: Superiority or Other; p = 0.005, ANCOVA — A priori threshold for statistical significance is p<0.05; Results obtained from ANCOVA with treatment, baseline and center in the model; LS mean treatment diff from placebo = -0.48, 95% CI 2-sided [-0.8 to -0.1]

4. Secondary Outcome: Change From Baseline in AM and PM Subject-reported Reflective Ocular Symptom Score Over the 2-week Treatment Period
Description: Participants recorded the severity of their ocular symptoms (Itching/burning eyes, tearing/watering eyes, and redness of eyes) over the past 12 hours (prior to the assessment) twice daily (AM and PM) using the following scale:
  0=absent (no sign/symptom present); 1=mild (sign/symptom present, easily tolerated); 2=moderate (definite awareness of sign/symptom, bothersome but tolerable); 3=severe (sign/symptoms hard to tolerate, interfere with daily activities).
  The total ocular symptom score ranges from 0 to 9 (worst symptoms). A negative change from baseline score indicates improvement.
Time Frame: Baseline (Days -3 to 0), and Days 1-15
Population: Intent to treat population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BDP HFA 320 µg/Day | Placebo
Number analyzed (Participants) | 167 | 171
units on a scale | -1.3 (0.13) | -0.7 (0.12)
Statistical Analysis 1: Comparison: BDP HFA 320 µg/Day vs Placebo; Test type: Superiority or Other; p = 0.002, ANCOVA — A priori threshold for statistical significance is p<0.05; [statistical method as in outcome 2, analysis 1]; LS mean treatment diff from placebo = -0.56, 95% CI 2-sided [-0.9 to -0.2]

ADVERSE EVENTS:
Arm/Group | BDP HFA 320 µg/Day | Placebo
Serious Adverse Events (participants affected / at risk) | 1/167 | 0/171
Other Adverse Events (participants affected / at risk) | 11/167 | 10/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BDP HFA 320 µg/Day (N=167) | Placebo (N=171)
Hypertensive crisis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BDP HFA 320 µg/Day (N=167) | Placebo (N=171)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 11 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.